CLINICAL TRIAL: NCT01483352
Title: Evaluation of Accu-Chek DiaPort, a Port System for Continuous Intraperitoneal Insulin Infusion, in Patients With Type I Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001211
Record Dates: First submitted 2011-11-15; First posted 2011-12-01 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- Single Arm (Experimental): Participants were implanted with Accu-Chek DiaPort with Infusion Set connected to an Accu-Chek Insulin Pump to perform continuous intraperitoneal insulin delivery.
  Interventions: Device: Accu-Chek DiaPort

INTERVENTIONS:
Device: Accu-Chek DiaPort

SUMMARY:
The Accu-Chek DiaPort system enables continuous intraperitoneal insulin infusion (CIPII): that is, infusion of insulin into the peritoneal cavity using an Accu-Chek insulin pump and an infusion set. The Accu-Chek DiaPort consists of a metal body with a catheter that is placed in the abdomen. The opening of the port is raised above the surface of the skin about 5 millimeters, while a flower-shaped plate is placed under the skin, providing stability for the port. The port has been designed for those diabetics who cannot benefit fully from subcutaneous insulin infusion. The primary objective of the study is to assess the suitability of Accu-Chek DiaPort to perform continuous intraperitoneal insulin delivery. The data collection focuses on the condition of tissue around the port after the implantation, possible peritoneal reactions to the port system, and the peritoneal delivery of insulin. Secondary objectives are the assessments of therapeutic performance and successful implementation of design requirements. In total 12 Patients will participate in this open, mono-centre, single-arm, interventional clinical trial. The study lasts 9 months (without run in period of 3 to 1 week) separated in two parts. Phase I last 12 weeks. Phase II last 6 month until the end of the study. During the study, seven visits are planned. The screening visit can take place up to 3 weeks before study start. At the implantation visit which can last up to 5 days the port will be implanted. After the implantation insulin therapy will be adjusted for CIPII and the patients will be trained for handling and daily care of the Accu-Chek DiaPort system. To check the functionality of the system, the first control visit will take place 2 weeks and the second control visit 6 weeks after the implantation. At the week 12 visit, the most important parameters will be collected for the phase I report. The following visits take place 6 and 9 months after the implantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >= 18 years of age at the time of the screening visit
* Type 1 diabetes mellitus
* On CSII therapy for at least 6 months prior to the screening visit
* Has been unsuccessfully treated with standard subcutaneous insulin therapy including CSII therapy, as defined by frequent (defined as handicapping in daily life) or severe (needing help from a third party) hypoglycemia and/or HbA1c above 8.5%, and/or other medical indication for CIPII therapy
* Presence of at least one of the following indications for CIPII therapy: - Frequent (defined as handicapping daily life) hypoglycemia during CSII therapy - Severe hypoglycemia (needing help from a third party) during CSII therapy - HbA1c above 8.5% during CSII therapy - Hypoglycemia unawareness during CSII therapy - Real subcutaneous insulin resistance - Insulin-induced lipoatrophy - Insulin-associated lipohypertrophy not controlled by site rotation - Other skin disorders interfering with the subcutaneous route of administration - Marked fluctuations of glucose levels and insulin requirements during CSII therapy- History of allergies to materials required for subcutaneous insulin therapy
* Performs usually self-management of blood glucose at least 4 times per day
* Willing to adhere to the study visit schedule and motivated to undergo the therapy

Exclusion Criteria:

* Presence of marked peritoneal adhesions or scarring after abdominal surgery
* Disorders of the gastrointestinal tract, respectively the digestive system potentially interfering with the intraperitoneal route of administration (e.g. presence of marked peritoneal adhesions, or colonic disease)
* Known high levels of anti-insulin antibodies
* History of allergy to materials used for the Accu-Chek DiaPort (titanium, polyethylene)
* Severely impaired immune response
* Uses systemic oral or inhaled steroids for > 14 days within the last 3 months
* Pregnant or lactating women, or women currently planning a pregnancy
* Previous history of severe chronic liver disease defined as signs of portal hypertension and/or Quick's value below 50% in spite of vitamin K administration
* Subject is treated for malignancy (chemotherapy, radiation or other treatment) (self-reported)
* Positive for HIV infection
* Is under CAPD treatment
* Suffers from severe eating disorders like bulimia or anorexia
* Alcohol or drug abuse
* Serious psychological disorders like schizophrenia, depression, Münchhausen's syndrome etc.
* Presence of known or suspected infections, bacteremia, septicemia or peritonitis
* Participation in a clinical trial (medicinal, medical device) within the last 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Holzer, Study Director — Roche Diabetes Care AG
Locations (1):
- Bad Heilbrunn, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Accu-Chek DiaPort: Participants were implanted with Accu-Chek® DiaPort with Infusion set connected to an Accu-Check Insulin Pump to perform continuous intraperitoneal insulin delivery.
Period: Overall Study
Arm/Group | Accu-Chek DiaPort
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received the implant were included in analysis.
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Suitability of the Device - Overall Suitability Score
Description: Suitability of the device was assessed by the investigator using a questionnaire that determined the following: 1) condition of the tissue around the port: tight connection between port and skin (mechanical stability, dislocation of port, signs of redness/swelling, infection, or pain), 2) peritoneal reactions (persistent dull pain due to catheter, signs of infection/allergic reaction) and ability to deliver insulin intraperitonally at every visit after implantation. Suitability score was determined using participant's responses to a questionnaire where 1 equals (=) no problem, 2=minor/negligible problems, 3=some/noticeable problems, 4=major/cumbersome and 5=severe/almost unbearable problems. Each question was scored and an average across the questions was determined as an overall score. The scores ranged from 1 (not at all suitable) to 5 (completely suitable).
Time Frame: Week 12
Population: All participants who received the implant were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
units on a scale | 2.00 (0.74)

2. Primary Outcome: Percentage of Participants With Problems Involving the Tight Connection Between Port and Skin
Description: Mechanical stability of the device was determined by the stability of the ingrowth surrounding the port as determined by the physician. The ingrowth problems are categorized as follows: Category 1= complete stable Ingrowth, 2= Ingrowth working with negligible problems, 3= Ingrowth working with some problems, 4= Ingrowth working with major problems and 5= Ingrowth resulting in almost non-functional port. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: All participants were included in the study; number (n)= number of participants analyzed for the given parameter at the specified timepoint
Measure: Number; unit: percentage of partcipants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of partcipants
  Category 1, Week 2 (n=12) | 33
  Category 2, Week 2 (n=12) | 50
  Category 3, Week 2 (n=12) | 17
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 75
  Category 2, Week 12 (n=12) | 25
  Category 3, Week 12 (n=12) | 0
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 36
  Category 2, Month 6 (n=11) | 55
  Category 3, Month 6 (n=11) | 9
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 55
  Category 2, Month 9 (n=11) | 46
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 70
  Category 2, Month 12 (n=10) | 30
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 64
  Category 2, Month 15 (n=11) | 27
  Category 3, Month 15 (n=11) | 9
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

3. Primary Outcome: Percentage of Participants With Dislocation of Port
Description: Position of the port was determined by the physician and was categorized as follows: Category 1= No dislocation; 2= Minimal dislocation; 3= Clearly visible dislocation, with minimal impairment of function; 4= Dislocation impairs functions; 5= Dislocation results in disabling functions. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: All participants were included in the analysis; n= number of participants analyzed for the given parameter at the specified timepoint
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 100
  Category 2, Week 2 (n=12) | 0
  Category 3, Week 2 (n=12) | 0
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 67
  Category 2, Week 12 (n=12) | 25
  Category 3, Week 12 (n=12) | 8
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 73
  Category 2, Month 6 (n=11) | 27
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 82
  Category 2, Month 9 (n=11) | 18
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 80
  Category 2, Month 12 (n=10) | 20
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 82
  Category 2, Month 15 (n=11) | 9
  Category 3, Month 15 (n=11) | 9
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

4. Primary Outcome: Percentage of Participants With Signs of Redness/Swelling in the Tissue Around the Port
Description: Signs of Redness/Swelling was determined by the physician and was categorized as follows: Category 1= None; 2= Minor, negligible; 3= Some, noticeable; 4= Major; 5= Severe. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 50
  Category 2, Week 2 (n=12) | 33
  Category 3, Week 2 (n=12) | 17
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 67
  Category 2, Week 12 (n=12) | 25
  Category 3, Week 12 (n=12) | 8
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 55
  Category 2, Month 6 (n=11) | 36
  Category 3, Month 6 (n=11) | 9
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 64
  Category 2, Month 9 (n=11) | 27
  Category 3, Month 9 (n=11) | 9
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 60
  Category 2, Month 12 (n=10) | 40
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 100
  Category 2, Month 15 (n=11) | 0
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

5. Primary Outcome: Percentage of Participants With Signs of Infection in the Tissue Around the Port
Description: Signs of infection were determined by the physician and categorized as follows : Category 1= None; 2= Minor, negligible; 3= Some, noticeable 4= Major; 5= Severe. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 75
  Category 2, Week 2 (n=12) | 8
  Category 3, Week 2 (n=12) | 17
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 83
  Category 2, Week 12 (n=12) | 17
  Category 3, Week 12 (n=12) | 0
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 100
  Category 2, Month 6 (n=11) | 0
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 91
  Category 2, Month 9 (n=11) | 9
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 90
  Category 2, Month 12 (n=10) | 10
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 64
  Category 2, Month 15 (n=11) | 36
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

6. Primary Outcome: Percentage of Participants With Signs of Pain in the Tissue Around the Port
Description: Signs of pain was determined from the participant questionnaire which was categorized as follows: category 1= No pain; 2= Minor, negligible; 3= Some, noticeable; 4= Major, cumbersome; 5=Severe, almost unbearable. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 83
  Category 2, Week 2 (n=12) | 17
  Category 3, Week 2 (n=12) | 0
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 100
  Category 2, Week 12 (n=12) | 0
  Category 3, Week 12 (n=12) | 0
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 100
  Category 2, Month 6 (n=11) | 0
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 91
  Category 2, Month 9 (n=11) | 9
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 80
  Category 2, Month 12 (n=10) | 20
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 100
  Category 2, Month 15 (n=11) | 0
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

7. Primary Outcome: Percentage of Participants With Persistent Dull Pain Due to Catheter
Description: Pain due to catheter was determined by a participant questionnaire and categorized as follows: Category 1= No pain; 2= Minor, negligible; 3= Some, noticeable; 4= Major, cumbersome; 5= Severe, almost unbearable. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 83
  Category 2, Week 2 (n=12) | 17
  Category 3, Week 2 (n=12) | 0
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 100
  Category 2, Week 12 (n=12) | 0
  Category 3, Week 12 (n=12) | 0
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 91
  Category 2, Month 6 (n=11) | 9
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 82
  Category 2, Month 9 (n=11) | 9
  Category 3, Month 9 (n=11) | 9
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 70
  Category 2, Month 12 (n=10) | 30
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5 Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 100
  Category 2, Month 15 (n=11) | 0
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

8. Primary Outcome: Percentage of Participants With Signs of Infection/Allergic Reaction at the Site of Implant
Description: Signs of infection/allergic reaction at the site of implant was determined by the physician and categorized as follows: 1= No problems; 2= Minor problems; 3= Some problems; 4= Major problems and/or replacement of catheter necessary; 5= Severe problems and/or explanation of port necessary. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 83
  Category 2, Week 2 (n=12) | 17
  Category 3, Week 2 (n=12) | 0
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 92
  Category 2, Week 12 (n=12) | 8
  Category 3, Week 12 (n=12) | 0
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 100
  Category 2, Month 6 (n=11) | 0
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 0
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 100
  Category 2, Month 9 (n=11) | 0
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 0
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 100
  Category 2, Month 12 (n=10) | 0
  Category 3, Month 12 (n=10) | 0
  Category 4, Month 12 (n=10) | 0
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 100
  Category 2, Month 15 (n=11) | 0
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 0
  Category 5, Month 15 (n=11) | 0

9. Primary Outcome: Percentage of Participants Categorized by Ability of the Port to Deliver Insulin Intraperitonally
Description: Problems in ability to deliver insulin intraperitoneally was determined by the physician and categorized as follows: 1= No problems; 2= Minor problems; 3= Some problems; 4= Major problems and/or replacement of catheter necessary; 5= Severe problems and/or explanation of port necessary. The percentage of participants in each category for the specified time point is presented.
Time Frame: Weeks 2 and 12 and Months 6, 9, 12 and 15
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Category 1, Week 2 (n=12) | 100
  Category 2, Week 2 (n=12) | 0
  Category 3, Week 2 (n=12) | 0
  Category 4, Week 2 (n=12) | 0
  Category 5, Week 2 (n=12) | 0
  Category 1, Week 12 (n=12) | 50
  Category 2, Week 12 (n=12) | 42
  Category 3, Week 12 (n=12) | 8
  Category 4, Week 12 (n=12) | 0
  Category 5, Week 12 (n=12) | 0
  Category 1, Month 6 (n=11) | 64
  Category 2, Month 6 (n=11) | 9
  Category 3, Month 6 (n=11) | 0
  Category 4, Month 6 (n=11) | 27
  Category 5, Month 6 (n=11) | 0
  Category 1, Month 9 (n=11) | 91
  Category 2, Month 9 (n=11) | 0
  Category 3, Month 9 (n=11) | 0
  Category 4, Month 9 (n=11) | 9
  Category 5, Month 9 (n=11) | 0
  Category 1, Month 12 (n=10) | 70
  Category 2, Month 12 (n=10) | 0
  Category 3, Month 12 (n=10) | 10
  Category 4, Month 12 (n=10) | 20
  Category 5, Month 12 (n=10) | 0
  Category 1, Month 15 (n=11) | 55
  Category 2, Month 15 (n=11) | 0
  Category 3, Month 15 (n=11) | 0
  Category 4, Month 15 (n=11) | 45
  Category 5, Month 15 (n=11) | 0

10. Secondary Outcome: Insulin Doses Dispensed From Insulin Pump
Description: Total insulin dose (in international units per milliliter [IU/mL]) from pump was measured per day as mean per day measured over 7 days.
Time Frame: Screening, Week 12 and Months 6, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
IU/mL
  Daily insulin dose - Screening (n=12) | 49.3 (53.2)
  Daily insulin dose - Week 12 (n=12) | 45.2 (30.1)
  Daily insulin dose - Month 6 (n=11) | 43.8 (32.7)
  Daily insulin dose - Month 9 (n=11) | 43.8 (36.4)
  Daily insulin dose - Month 12 (n=10) | 40.8 (34.5)
  Daily basal insulin dose - Screening (n=12) | 9.6 (4.8)
  Daily basal insulin dose - Week 12 (n=12) | 11.1 (5.1)
  Daily basal insulin dose - Month 6 (n=11) | 9.9 (4.5)
  Daily basal insulin dose - Month 9 (n=11) | 10.1 (4.5)
  Daily basal insulin dose - Month 12 (n=10) | 9.3 (4.6)
  Daily bolus insulin dose - Screening (n=12) | 39.6 (49.3)
  Daily bolus insulin dose - Week 12 (n=12) | 34.1 (26.9)
  Daily bolus insulin dose - Month 6 (n=11) | 33.8 (29.6)
  Daily bolus insulin dose - Month 9 (n=11) | 33.7 (33.2)
  Daily bolus insulin dose - Month 12 (n=10) | 31.6 (31.0)

11. Secondary Outcome: Hemoglobin A1c Levels
Description: Glycated hemoglobin (HbA1c) is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. HbA1c levels are a measure of glycemic control.
Time Frame: Screening, Week 12 and Months 6, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of glycated hemoglobin
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percent of glycated hemoglobin
  Screening (n=12) | 8.99 (1.13)
  Week 12 (n=12) | 7.99 (0.97)
  Month 6 (n=11) | 7.57 (0.64)
  Month 9 (n=11) | 7.73 (1.01)
  Month 12 (n=10) | 8.38 (1.15)

12. Secondary Outcome: Self Monitored Blood Glucose Levels
Description: Participants monitored glucose levels on a daily basis and recorded for evaluation. Glucose levels are measured as milligrams per deciliter (mg/dL)
Time Frame: Screening, Week 12 and Months 6, 9 and 12
Population: All participants were included in analysis; n= number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
mg/dL
  Screening (n=12) | 185.1 (33.0)
  Week 12 (n=12) | 176.6 (31.1)
  Month 6 (n=11) | 164.1 (30.6)
  Month 9 (n=11) | 174.7 (44.2)
  Month 12 (n=10) | 184.6 (36.6)

13. Secondary Outcome: Continuous Glucose Measurement (CGM) - Glucose Levels
Description: CGM measurements were performed using a diurnal CGM sensor and group means were calculated over 10 minute periods of the CGM measurements.
Time Frame: Screening, Week 12 and 6 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
mg/dL
  Screening (n=12) | 200.7 (39.6)
  Week 12 (n=12) | 174.3 (20.3)
  Month 6 (n=11) | 173.4 (24.9)

14. Secondary Outcome: Glycemic Variability: Percent Coefficient of Variation in Blood Glucose
Description: Both self monitored (SMBG) and continuous (CGM) glucose measurements were used to determine the coefficient of variation in blood glucose. CGM data are only evaluated for a 1 week time period and are no direct comparison to the SMBG that reflect the full time frame between visits.
Time Frame: Screening, Week 12 and Months 6, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of mean glucose value
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percent of mean glucose value
  SMBG - Screening (n=12) | 45.1 (9.8)
  SMBG - Week 12 (n=12) | 38.4 (5.9)
  SMBG - Month 6 (n=11) | 41.7 (9.4)
  SMBG - Month 9 (n=11) | 38.5 (7.2)
  SMBG - Month 12 (n=10) | 38.8 (7.1)
  CGM - Screening (n=12) | 40.3 (8.5)
  CGM - Week 12 (n=12) | 37.8 (9.0)
  CGM - Month 6 (n=11) | 38.2 (9.8)

15. Secondary Outcome: Percentage of Participants Achieving Target Glucose Levels
Description: Target glucose values were 70-180 mg/dL. Participants with glucose levels below 70 mg/dL were considered to be under target and those above 180 mg/dL were considered over target. The mean of Glucose-Measurements at the visit date was calculated as follows: a variable was created for each category ("within target [70-180 mg]", "below target" and "above target") that tells if the value lies within this category. Then the percentage per participant and visit was calculated. The mean represents the mean of these percentages per participant at the visit.
Time Frame: Screening, Week 12 and 6 Months
Population: All participants were included in the study; n= number of participants analyzed for the given parameter at the specified timepoint
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Within target range - Screening (n=12) | 44.6 (14.4)
  Within target range - Week 12 (n=12) | 56.5 (12.0)
  Within target range - Month 6 (n=11) | 58.3 (13.1)
  Above target range - Screening (n=12) | 52.6 (15.5)
  Above target range - Week 12 (n=12) | 39.9 (11.7)
  Above target range - Month 6 (n=11) | 37.8 (13.5)
  Below target range - Screening (n=12) | 2.9 (2.8)
  Below target range - Week 12 (n=12) | 3.6 (3.7)
  Below target range - Month 6 (n=11) | 3.8 (4.8)

16. Secondary Outcome: Design Validation Participant Questionnaire - Percentage of Participants With a Positive Response
Description: The participant questionnaire consisted of two parts including description of routine operations, followed by 23 questions used to determine the following: percentage of participants needing consultation of instructions for use of fixation disc or infusion set; percentage of participants with pain after implantation, percentage of participants with moderate pain during 4 to 6 days after implantation, moderate pain for 7 days or more; percentage of participants with temporal disconnection from infusion set; percentage of participants with use of handling aid for temporal storage; percentage of participants with a reason for temporal disconnection of infusion set from port either sex, shower, or sport; percentage of participants changing fixation disc ≥3 days or infusion set ≥4 days and the cartridge, and percentage of participants cleaning the skin around the port daily, every second day, or every third to fifth day, either with saline during healing or with alcohol after healing.
Time Frame: Week 12
Population: All participants were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Accu-Chek DiaPort
Number analyzed (Participants) | 12
percentage of participants
  Needing Instruction for Fixation disc | 92
  Needing Instruction for Infusion set | 92
  With Pain after implantation | 75
  Moderate pain after implantation during 4 - 6 days | 17
  Moderate pain after implantation 7 days or more | 17
  Disconnection of infusion set from port-daily | 33
  Disconnection of infusion set from port-never | 33
  Stopped pump during temporal disconnection | 17
  Used handling aid for temporal storage | 83
  Reason for temporal disconnection-sex | 33
  Reason for temporal disconnection-shower | 83
  Reason for temporal disconnection-sport | 17
  Changed fixation disc after ≥3 days | 75
  Changed infusion set after ≥4 days | 83
  Changed cartride and infusion set simultaneously | 92
  Changed fixation disc and cartridge simultaneously | 55
  Cleaned skin around port-daily | 50
  Cleaned skin around port-every second day | 17
  Cleaned skin around port-3rd to 5th day | 17
  Cleaned skin around port-with saline | 58
  Cleaned skin around port-with alcohol | 50

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of implantation until the end of study.
Arm/Group | Accu-Chek DiaPort
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accu-Chek DiaPort (N=12)
Diaport replacement (Injury, poisoning and procedural complications) | 1
Complete catheter occlusion (Injury, poisoning and procedural complications) | 1
Catheter replacement (Injury, poisoning and procedural complications) | 2
Over growth of abdominal catheter (Injury, poisoning and procedural complications) | 1
Symptomatic hypoglycemia (Endocrine disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Diabetic ketoacidosis (Endocrine disorders) | 1
Instable blood sugar (Endocrine disorders) | 1
Coronary bypass surgery (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accu-Chek DiaPort (N=12)
Chronic ischaemic heart disease (Cardiac disorders) | 1
Chronic lower respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1
Complications of other internal prosthetic devices, implants and grafts (Surgical and medical procedures) | 7
Disease of pancreas, unspecified (Gastrointestinal disorders) | 1
Diseases of oesophagus, stomach and duodenum (Gastrointestinal disorders) | 1
Disorders of lipoprotein metabolism and other lipidaemias (Metabolism and nutrition disorders) | 1
Dorsalgia, unspecified (Musculoskeletal and connective tissue disorders) | 1
Essential (primary) hypertension (Vascular disorders) | 2
Functional diarrhea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Hypertensive disease (Vascular disorders) | 1
Insulin-dependent diabetes mellitus (Metabolism and nutrition disorders) | 7
Insulin-dependent diabetes mellitus with renal complications (Metabolism and nutrition disorders) | 2
Mental and behavioural disorders (Psychiatric disorders) | 2
Metabolic disorders (Metabolism and nutrition disorders) | 1
Other and unspecified medical devices associated with adverse incidents (Surgical and medical procedures) | 10
Other diseases of intestines (Gastrointestinal disorders) | 1
Other diseases of upper respiratory tract (Respiratory, thoracic and mediastinal disorders) | 1
Other diseases of urinary system (Renal and urinary disorders) | 1
Other soft tissue disorders, not elsewhere classified (Musculoskeletal and connective tissue disorders) | 1
Pain localized to upper abdomen (Gastrointestinal disorders) | 1
Presents of coronary angioplasty implant and graft (Surgical and medical procedures) | 1
Scar conditions and fibrosis of skin (Skin and subcutaneous tissue disorders) | 1
Superficial injury of unspecified body region (Injury, poisoning and procedural complications) | 1
Symptoms and signs involving the digestive system and abdomen (Gastrointestinal disorders) | 1
Urinary tract infection, site not specified (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.